2020N435833 00

The GlaxoSmithKline group of companies

207863

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK3732394 in Healthy Participants |
|---|---|---|
| <b>Compound Number</b> | : | GSK3732394 |
| <b>Effective Date</b> | : | 04-MAY-2020 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Synoptic Clinical Study Report for Protocol 207863.
- This RAP is intended to describe the safety, tolerability, pharmacokinetic, and pharmacodynamic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Part 1 (Single Ascending Dose) Statistical Analysis Complete (SAC) deliverable. Due to early termination of the study only the first 3 cohorts were completed. This document will only include the reporting plan for subjects enrolled in the study.
- Only the primary and secondary endpoints are to be analysed due to the early termination.

#### Author(s):

| Lead | Date |
|---|---|
| Principal Statistician (Infectious Diseases, Biostatistics) | 30-APR-2020 |
| Co-Author PPD 30-APR-2020 Manager (Clinical Pharmacology Modelling Simulation) | |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

2020N435833\_00

The GlaxoSmithKline group of companies

207863

# **RAP Team Review Confirmations (Method: E-mail)**

| Approver | Date |
|---|---|
| PPD (L. C. J. D. D. L. J. | 30-APR-2020 |
| Principal Programmer (Infectious Disease, Biostatistics) | |
| PPD | |
| Clinical Science Director (ViiV Healthcare, Clinical Development) | 30-APR-2020 |

# Clinical Statistics and Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | |
|-------------------------------|-------------------------|
| PPD | |
| Statistics Leader (I | D, Clinical Statistics) |
| PPD | |
| Programming Dire Programming) | ctor (ID, Clinical |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRODUCT | ION | 6 |
| 2. | SUMMARY O | F KEY PROTOCOL INFORMATION | 7 |
| ۷. | | ges to the Protocol Defined Statistical Analysis Plan | |
| | | Objective(s) and Endpoint(s) | |
| | , | Design | |
| | | ical Analyses | |
| 3. | PI ANNED AN | VALYSES | 11 |
| ٠. | | n Analyses | |
| | | Analyses | |
| 4. | ANALYSIS PO | OPULATIONS | 12 |
| ٠. | | col Deviations | |
| 5. | | TIONS FOR DATA ANALYSES AND DATA HANDLING NS | 10 |
| | | Treatment & Sub-group Display Descriptors | |
| | | ne Definitions | |
| | | Considerations for Data Analyses and Data Handling | 10 |
| | Conve | entions | 14 |
| 6. | STI IDV DODI | JLATION ANALYSES | 15 |
| 0. | | iew of Planned Study Population Analyses | |
| | O.T. OVERV | ow of Flammod Stady Fopulation / than your | |
| 7. | | LYSES | |
| | | se Events Analyses | |
| | | al Laboratory Analyses | |
| | | Safety Analyses | |
| | 7.3.1. | <b>0</b> | |
| | 7.3.2. | <b>.</b> | |
| | 7.3.3. | Liver Events | 18 |
| 8. | PHARMACO | KINETIC ANALYSES | 19 |
| | 8.1. Pharm | nacokinetic Parameter Definitions and Summaries | |
| | 8.1.1. | Endpoint / Variables | |
| | | 8.1.1.1. Drug Concentration Measures | |
| | | 8.1.1.2. Derived Pharmacokinetic Parameters | |
| | 8.1.2. | Summary Measure | |
| | 8.1.3. | Population of Interest | |
| | 8.1.4. | Strategy for Intercurrent (Post-Randomization) Events | |
| | 8.1.5. | Statistical Analyses / Methods | |
| | | ical Analysis of derived PK Parameters | |
| | 8.2.1. | Endpoint / Variables | |
| | 8.2.2. | Summary Measure | |
| | 8.2.3. | Population of Interest | |
| | 8.2.4.<br>8.2.5 | Strategy for Intercurrent (Post-Randomization) Events | 21<br>21 |

# 2020N435833\_00

# CONFIDENTIAL

| 207 | 863 |
|-----|-----|
|-----|-----|

| | | | 8.2.5.1. | Statistical Methodology Specification | .21 |
|---|---|---|---|---|---|
| 9. | PHARI | MACODY | NAMIC AN | ALYSES | 23 |
| ٠. | 9.1. | | | Parameters and Summaries | |
| | 0.1. | 9.1.1. | | Variables | |
| | | 9.1.2. | | Measure | |
| | | 9.1.3. | | of Interest | |
| | | 9.1.4. | | or Intercurrent (Post-Randomization) Events | |
| | | 9.1.5. | | Analyses / Methods | |
| | | 0.1.0. | Otatiotical | , that you have the same the same that the same | |
| 10. | REFE | RENCES. | | | . 25 |
| 11 | ΔΡΡΕΙ | NDICES | | | 26 |
| | 11.1. | | | I Deviation Management and Definitions for Per | . 20 |
| | | | | | 26 |
| | 11.2. | | | le of Activities | |
| | 11.3. | | | ment Windows | |
| | 11.5. | | | of Assessment Windows for Analyses | |
| | 11.4. | | | Phases and Treatment Emergent Adverse | . 00 |
| | 11.4. | | | mases and Treatment Emergent Adverse | .34 |
| | | 11.4.1. | | ses | |
| | | | • | Study Phases for Concomitant Medication | |
| | | 11.4.2. | | Emergent Flag for Adverse Events | |
| | 11.5. | | | splay Standards & Handling Conventions | |
| | | 11.5.1. | | Process | |
| | | 11.5.2. | | Standards | |
| | | 11.5.3. | | Standards for Pharmacokinetic Data | |
| | 11.6. | | 6: Derived | I and Transformed Data | .37 |
| | | 11.6.1. | | | |
| | | 11.6.2. | | ulation | |
| | | 11.6.3. | | | |
| | | 11.6.4. | | kinetic | |
| | | 11.6.5. | | dynamic | |
| | 11.7. | | | ng Standards for Missing Data | |
| | | 11.7.1. | Premature | Withdrawals | 40 |
| | | | | of Missing Data | |
| | | | | Handling of Missing and Partial Dates | |
| | 11.8. | Annendix | | of Potential Clinical Importance | |
| | 11.0. | 11.8.1. | Laboratory | Values | 42 |
| | | 11.8.2. | | V44400 | |
| | 11.9. | Annendix | 9. Abbrev | ations & Trade Marks | 43 |
| | 11.0. | 11.9.1. | | ons | |
| | | 11.9.2. | | (\$ | |
| | 11 10 | | | Data Displays | |
| | 11.10. | | | ay Numbering | |
| | | | | es | |
| | | | | ulation Tables | |
| | | | | ples | |
| | | | | kinetic Tables | |
| | | | | kinetic Figures | |
| | | | | dynamic Tables | |
| | | 11.10.7. | i Haililaco | uynanno rabies | . JU |

| | CONFIDENTIAL | 2020N435833_00<br>207863 |
|----------|------------------|--------------------------|
| 11.10.8. | ICH Listings | 51 |
| | Non-ICH Listings | |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 207863:

| Revision Chronology: | | |
|---|---|---|
| Original Protocol,<br>DNG<br>2017N341355_00 | 11-APR-2019 | Original |
| Amendment 01, DNG 2017N341355_01 | 06-JUN-2019 | This amendment results from FDA "Study May Proceed" letter for IND Opening (Number 131394, Reference ID 4441322) dated 31-MAY-2019. FDA requested 9 clinical changes to the protocol. |
| Amendment 02, DNG 2017N341355_02 | 02-JUL-2019 | This amendment results from a consensus between the Sponsor and the Study Site, that a confirmation of CD4+ T-cell count and CD4 percent values in healthy individuals with values within the normal range at screening, to be unnecessary. The removal of this confirmatory test is not determined to have effect on the evaluation of participant safety by the Sponsor or Study Site. |
| Amendment 03, DNG 2017N341355_03 | 12-SEP-2019 | This amendment is based on 3 criteria. 1) Initial dose escalation data following completion of Cohort 1 indicated that Cohort 6 in the study design will be required. Flexible language to this affect has been removed. 2) Initial dose escalation data following completion of Cohort 1 indicate that anti-drug antibodies (ADA) have the potential to appear earlier than indicated pre-clinically. Day 7 and Day 10 collection of samples for ADAs have been added in Part 1 and for Day 8 in Part 2. 3) The previous consensus between the Sponsor and the Study Site on CD4+ T-cell count and CD4 percent values screening values under Amendment 02, requires further clarification. |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| <ul> <li>No changes or deviations<br/>specified in protocol amendment</li> <li>3.</li> </ul> | No Statistical Analysis or<br>outputs to be generated for<br>Part 2 (Multiple Ascending<br>Dose) or exploratory<br>objectives/endpoints | Study terminated prior to<br>multiple dosing |
| Full CSR | Synoptic CSR | Early study termination<br>during Part 1 for non-safety<br>reasons. |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the safety and tolerability of single and multiple doses of GSK3732394 in healthy participants. | GSK3732394 safety parameters: adverse events; post-baseline values and changes over time of clinical laboratory evaluations (haematology, clinical chemistry, urinalysis), vital signs, and ECG parameters from predose values |
| Secondary Objectives | Secondary Endpoints |
| To describe the pharmacokinetic<br>(PK) profile of single and multiple<br>doses of GSK3732394 in healthy<br>participants. | <ul> <li>Derived PK parameters for GSK3732394, as data allow: Part 1 (single dose): AUC<sub>(0-t)</sub>, AUC<sub>(0-∞)</sub>, C<sub>max</sub>, T<sub>max</sub>, t<sub>lag</sub>, C<sub>last</sub>, t<sub>last</sub>, t<sub>1/2</sub>,CL/F</li> <li>Part 2 (Repeated Once Weekly [QW] dosing): First week: AUC<sub>(0-t)</sub>, AUC<sub>(0-∞)</sub>, C<sub>max</sub>, t<sub>max</sub>, t<sub>lag</sub></li> <li>Last week: AUC<sub>(0-t)</sub>, C<sub>max</sub>, t<sub>max</sub>, C<sub>trough</sub>, t<sub>1/2</sub>, CL/F.</li> </ul> |
| To examine dose proportionality<br>following single and multiple doses<br>of GSK3732394, as data allow. | <ul> <li>PK linearity assessment using derived PK parameters, as data allow: Part 1 (single dose): AUC<sub>(0-∞)</sub>, C<sub>max</sub> </li> <li>Part 2 (Repeat QW dosing): AUC<sub>(0-τ)</sub>, C<sub>max</sub>, C<sub>τ</sub>.</li> </ul> |
| <ul> <li>To assess accumulation of<br/>GSK3732394 after multiple doses,<br/>as data allow.</li> <li>To characterise CD4 receptor<br/>occupancy (RO) profile of single<br/>and multiple doses of<br/>GSK3732394.</li> </ul> | <ul> <li>Accumulation indices for PK parameters assessed across first and last doses of multiple dosing, as data allow: RAUC<sub>(0-τ)</sub>, RC<sub>max</sub>, RC<sub>τ</sub>.</li> <li>Percent of CD4 RO.</li> </ul> |
| To investigate the relationship | C <sub>max</sub> , C <sub>trough</sub> , %RO |

| Objectives | Endpoints |
|---|---|
| between GSK3732394 exposures and CD4 RO. | |
| To characterise potential immunologic impact on, and immune responses to, healthy participants who receive a single or multiple dose(s) of GSK3732394. | <ul> <li>Change from baseline in CD3/CD4/CD8 and activated T-cell counts and percentages.</li> <li>Change from baseline in CD4 mean fluorescence intensity (MFI).</li> <li>Titers and incidence of anti-GSK3732394 antibodies.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To model the relationship between<br>GSK3732394 exposures and CD4<br>RO. | Estimating parameters descriptive of the relationship including Concentration resulting in 50% RO (EC50), as data allow. |
| To explore the correlation between<br>GSK3732394 exposure and<br>observed safety outcomes. | Occurrence of AEs /laboratory abnormalities and<br>corresponding plasma concentrations / doses of<br>GSK3732394. |
| To explore serum and urine<br>metabolite(s) investigations of<br>GSK3732394. | Identification of any compound-related degradants |

### 2.3. Study Design

#### Overview of Study Design and Key Features

#### Schematic:

| PART1 | SAD Cohort1 | SAD Cohort2 | SAD Cohort3 | SAD Cohort 4 | SAD Cohort 5 | SAD Cohort 6 <sup>1</sup> |
|---|---|---|---|---|---|---|
| (6 GSK3732394:2 PBO) | (n = 8) | (n = 8) | (n = 8) | (n = 8) | (n =8) | (n = 8) |
| Single SC Dose | 10mg | 40mg | 130mg | 350mg | 600mg | Up to 800mg or to |
| (C <sub>trough</sub> RO) | (<10%) | (≤25%) | (≤70%) | (≤90%) | (≤95%) | repeata prior dose |

| PART 2 | MAD Cohort1 | MAD Cohort 2 | MAD Cohort 3 |
|---|---|---|---|
| (6 GS K3732394 : 2 PBO) | (n = 8) | (n = 8) | (n = 8) |
| 4 Subcutaneous Doses (C <sub>bough</sub> RO) | 130mg | 400mg | 600mg |
| Administered Once Weekly (QW) | (<70%) | (≤90%) | (≤95%) |

<sup>1</sup> An additional cohort (6) of up to 800mg or to repeat a prior dose may be included.

Note: Doses shown in schematic are nominal and intended to demonstrate general concepts relating to factors of escalation as a base case. Dose escalation in Part 1 will be based on target receptor occupancy/exposure and governed by safety and PK stopping criteria. Transition to Part 2 will be after the completion of dosing and evaluation of SAD Cohort 4 participants and after the predicted exposure of the starting MAD dose is within that observed with SAD dosing – maximum predicted AUC, Cmax not exceeding the average maximum observed in evaluated SAD cohorts. (QW = once every week.).

# Design Features

- 2 Part, double-blind (sponsor-unblinded), randomized, placebo-controlled, single and multiple-ascending-dose study.
- In Part 1, a sufficient number of healthy adults will be screened to provide approximately 8 participants for randomization within each of the SAD dosing cohorts. Overall, up to approximately 48 participants will be included depending on the number of cohorts required.
- In Part 2, a sufficient number of healthy adults will be screened to provide approximately 8 participants for randomization within each of the 3 MAD dosing cohort. Overall, up to approximately 24 participants will be included depending on the number of cohorts required.

#### Dosing

- In Part 1, the proposed dosing schedule is designed to investigate SAD of GSK3732394 in healthy participants. All doses will be administered subcutaneously. The SAD portion of the study will be conducted in at least five, but no more than six, separate cohorts of approximately eight healthy adult participants each. Each of the participants in the SAD cohorts will receive a single dose of blinded GSK3732394 or blinded PBO (GSK3732394: PBO = 6:2, per their randomization assignment). Details of the starting dose and dose escalation can be found in Section 5.5.1 and Section 5.5.2, respectively, of the protocol. Dose escalation decisions, including the determination of subsequent doses in Part 1, will be determined by the Safety and Dose Escalation Committee (SDEC). See Section 5.5.5 of the protocol.
- In Part 2, the proposed dosing schedule is designed to investigate multiple ascending doses (MAD) of GSK3732394 in healthy participants administered weekly for a total of four doses. All doses will be administered subcutaneously.
- Part 2 consists of up to three ascending repeat-dose cohorts (MAD Cohorts 1, 2, and 3), each with approximately 8 participants (GSK3732394 : PBO = 6:2) who will receive four weekly doses of GSK3732394 or PBO on Days 1, 8, 15, and 22. Details of starting dose and dose escalations in Part 2 (MAD) can be

| Overview of St | udy Design and Key Features |
|---|---|
| | found in Section 5.5.3 of the protocol. |
| Time & | Refer to Appendix 2: Schedule of Activities |
| Treatment<br>Assignment | <ul> <li>In Part 1, participants will receive a single dose of GSK3732394 or PBO (6:2) on Day 1. Safety, PK and PD assessments will be performed at timepoints specified in the schedule of activity (SOA). Participants will remain in the clinic until the completion of the Day 14 procedures and will return to the clinic on Days 17, 21, and 24 for follow-up assessments, and an end-of-study evaluation on Day 28.</li> <li>In Part 2, participants will receive doses of GSK3732394 or PBO (6:2) given at anticipated weekly intervals. Participants will remain in the clinic until the completion of the Day 35 procedures and will return to the clinic on Days 39, 42 and 46 for follow-up assessments, and an end-of-study evaluation on Day 49. Duration of participation through follow-up may be longer if actual PK parameters differ significantly from predicted values (e.g. if half-life is significantly longer than the predicted); but will not exceed five half-lives.</li> </ul> |
| Interim<br>Analysis | No formal interim analyses (IA) are planned for this study. However, safety, tolerability, PK, and PD data will be reviewed before each dose escalation in Part 1 (single dose). Part 2 (report dose) and prior to MAD transition which will. |
| | Part 1 (single dose), Part 2 (repeat dose) and prior to MAD transition which will occur after at least the first 4 SAD cohorts. |

# 2.4. Statistical Analyses

The main purpose of this study is to assess the safety, tolerability, and pharmacokinetic/pharmacodynamic attributes of subcutaneous doses of GSK3732394 in healthy participants. No formal hypotheses will be tested. Results will be descriptive in nature. Statistical modelling on select pharmacokinetic parameters will be performed to estimate dose proportionality. Point estimates with 90% confidence intervals will be reported, as appropriate.

## 3. PLANNED ANALYSES

# 3.1. Interim Analyses

There will be no formal interim analysis; however, all preliminary safety, tolerability, and available PK/PD data will be reviewed internally prior to each dose escalation and prior to transitioning to MAD dosing. Dose escalation can only occur after the Safety and Dose Escalation Committee (SDEC) has found that the safety, PK/PD profiles are supportive to proceed with the evaluation of the next higher dose level. The details of internal review process to support dose-escalation are included in the SDEC charter document.

After each cohort, the data will be reviewed – the data consists of the PK, RO, relationship between PK and RO, and safety data. At each cohort dose review, a dose will be proposed that meets the RO requirements for the next dosing cohort. Non-compartmental analysis (NCA) PK analysis will be performed to obtain PK parameters.

Beginning with the second dose in Part 1 and each subsequent dose throughout the study, the Bayesian probability of any individual participant exceeding the  $C_{max}$  No Observed Adverse Effect Level (NOAEL) exposure of 93.9  $\mu$ g/mL (Protocol Section 5.5.1) at that dose will be calculated, using the accumulated PK data of participants receiving GSK3732394 among the previous cohorts. Observations on placebo will be excluded. This probability, together with safety and tolerability data of the preceding cohorts, will be used to help selection of the next dose. The Bayesian probability of exceeding the  $C_{max}$  threshold can be calculated for additional potential doses to aid in dose selection if necessary.

The Bayesian probability will be based on Whitehead's model shown below [Whitehead, 2001] using non-informative priors for the model parameters.  $v_i = \theta_1 + \theta_2 d_i + \varepsilon_i$ 

Where  $y_i$  is log-PK of i-th participant,  $d_i$  is the log-dose administered to i-th participant.  $\theta_1$  and  $\theta_2$  are population intercept and slope, respectively.  $\epsilon_i$  is the random error of the i-th participant.

For the prediction of the second dose in Part 1 and Part 2,  $\theta_2$  will be assumed to equal 1 (representing a dose proportionality assumption). This will allow for the estimation of the remaining parameters of the model using data from only one dose level.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants at the time of termination of the study have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.

- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Study Population</li> </ul> |
| Enrolled | All participants who passed screening and were randomized. | Study Population |
| | Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | |
| Safety | All participants who received at least 1 dose of study treatment. Participants will be analyzed according to the treatment they actually received. | <ul><li>Study Population</li><li>Safety</li></ul> |
| | Note: Participants who were not randomized but received at least one dose of study treatment should be listed. | |
| Pharmacokinetic | All participants in the Safety population who had at least | • PK |
| (PK) | 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). | • PD |

Refer to **Section 11.10**: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF (ClinBase).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptors | | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code Description | | Description | Order in TLF |
| Part 1 | | | |
| А | GSK3732394 Single dose level 1 | GSK3732394 Single Dose<br>10 mg | 1 |
| В | GSK3732394 Single dose level 2 | GSK3732394 Single Dose<br>20 mg | 2 |
| С | GSK3732394 Single dose level 3 | GSK3732394 Single Dose<br>80 mg | 3 |
| Р | Placebo | Single Dose Placebo | 4 |

#### **NOTES:**

• Order represents treatments being presented in TLF, as appropriate.

#### 5.2. Baseline Definitions

For all endpoints the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. The Table below illustrates this rule for the planned Study Assessments. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments Considered as Baseline | | | Baseline to use in |
|---|---|---|---|---|
| | Screening | creening Day -1 Day 1 (Pre-Dose) | | Data Display |
| Part 1 | | | | |
| Vital Signs, ECG | X | | X | Day 1 (Pre-Dose) |
| PK sample, PD<br>Sample | | | X | Day 1 (Pre-Dose) |
| Lab Assessments | Х | Х | | Day -1 |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

2020N435833\_00 207863

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 11.3 | Appendix 3: Assessment Windows |
| 11.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 11.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 11.6 | Appendix 6: Derived and Transformed Data |
| 11.7 | Appendix 7: Reporting Standards for Missing Data |
| 11.8 | Appendix 8: Values of Potential Clinical Importance |

2020N435833\_00

207863

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, concomitant medications, and exposure will be based on GSK Core Data Standards. Details of the planned displays are presented in Section 11.10: List of Data Displays.

7. SAFETY ANALYSES

The safety analyses will be based on the safety population, unless otherwise specified. All details of the planned displays are provided in Section 11.10: List of Data Displays. Unless otherwise specified, endpoints/variables will be summarized using descriptive statistics and listed.

### 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Section 11.10: List of Data Displays.

AEs will be coded to the preferred term (PT) level using the Medical Dictionary for Regulatory Affairs (MedDRA) V22.1. AEs will be graded by the investigator according to the Division of AIDS (DAIDS) Criteria Version 2.1.

Injection site reactions will be reported as adverse events and included in the adverse events displays. Multiple symptoms of injection site reactions will be reported as separate adverse events for each reported symptom.

A summary of non-serious AEs that occurred in strictly 5% of the participants or above will be provided (even with the limited sample size of the study, no rounding for the percentage will be used in terms of 5% threshold).

A summary of number and percentage of participants with any adverse event by maximum grade will be produced. AEs will be sorted by PT in descending order of total incidence. The summary will use the following algorithms for counting the participant:

- Preferred term row: Participants experiencing the same AE preferred term several times with different grades will only be counted once with the maximum grade.
- Any event row: Each participant with at least one adverse event will be counted only once at the maximum grade no matter how many events they have.

The following listings will be provided:

- All adverse events
- Subject Numbers for Individual AEs

# 7.2. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests (with lymphocyte subset [CD4/CD8/CD3]), Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Section 11.10: List of Data Displays. Haematology, clinical chemistry and urinalysis parameters collected are listed below:

| Laboratory | Parameters | | | |
|---|---|---|---|---|
| Assessments | | | | |
| Hematology | Platelet Count<br>RBC Count<br>Hemoglobin<br>Hematocrit | RBC Indices:<br>MCV<br>MCH<br>%Reticulocytes | WBC count with Differential: Neutrophils Lymphocytes Monocytes Eosinophils Basophils | Lymphocyte Phenotype Absolute number and Percent of: CD3+ CD4+ CD8+ |
| Clinical Chemistry | BUN | Potassium | Aspartate Aminotransferase (AST)/ Serum Glutamic-Oxaloacetic Transaminase (SGOT) | Total and direct bilirubin |
| | Creatinine | Sodium | Alanine Aminotransferase (ALT)/ Serum Glutamic-Pyruvic Transaminase (SGPT) | Total Protein |
| | Glucose | Calcium | Alkaline phosphatase | Amylase |
| | Lipase | | | |
| Routine Urinalysis | <ul> <li>Specific gravity</li> <li>pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase by dipstick</li> <li>Microscopic examination (if blood or protein is abnormal)</li> </ul> | | | |
| Other Screening<br>Tests | <ul> <li>Follicle-stimulating hormone and estradiol (as needed in women of non-childbearing potential only)</li> <li>Serum alcohol and urine drug screen (to include at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines)]</li> <li>Serum human chorionic gonadotropin (hCG) pregnancy test (as needed)<sup>2</sup></li> <li>Serology [(HIV antibody, hepatitis B surface antigen [HBsAg], and hepatitis C virus antibody)]</li> <li>Creatinine clearance (CrCL) for GFR estimation</li> <li>The results of each test must be entered into the CRF.</li> </ul> | | | |

Laboratory toxicity grading will follow DAIDS grading criteria. Parexel data management will apply the grading in the SDTM dataset.

# 7.3. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Section 11.10: List of Data Displays.

#### 7.3.1. Vital Signs

Vital sign values and change from baseline will be summarized. In addition, the number of subjects with worst case vital sign results relative to potential clinical importance (PCI) criteria post-baseline relative to baseline will be summarized by test and category.

207863 | Statistical Analysis Plan RAP 04 May 2020 | TMF-1766872 | 2.0

CONFIDENTIAL

2020N435833\_00 207863

# 7.3.2. Electrocardiograms

A summary of the number and percentage of subjects of all ECG findings will be displayed by treatment. Additionally, summary statistics of ECG values and change from baseline in ECG values will be presented.

#### 7.3.3. Liver Events

The number of events does not support a summary. Liver monitoring/stopping event reporting will therefore only be listed for participants with liver events. In addition, listings will be produced for medical conditions and substance use for participants with liver events.

## 8. PHARMACOKINETIC ANALYSES

All PK analyses planned for the study are either part of the secondary or exploratory objectives. Due to study termination, only secondary PK analyses will be reported. The PK analyses will be based on the PK population, unless otherwise specified.

#### 8.1. Pharmacokinetic Parameter Definitions and Summaries

## 8.1.1. Endpoint / Variables

#### 8.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 11.5.3 Reporting Standards for Pharmacokinetic)

#### 8.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin version 8.0. All calculations of non-compartmental parameters for the final analysis will be based on planned sampling times. Planned sampling times will be used due to early termination of the study and the frequency of PK sampling times in Part 1. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| $C_{max}$ | Maximum observed concentration, determined directly from the concentration-time data. |
| t <sub>max</sub> | Time to reach C <sub>max</sub> , determined directly from the concentration-time data. |
| t <sub>lag</sub> | Lag time before observation of drug concentrations (after single dose only) |
| C <sub>last</sub> | last observable concentration |
| t <sub>last</sub> | time of last quantifiable concentration |
| t <sub>1/2</sub> | Apparent terminal phase half-life calculated as $t_{1/2} = \frac{\ln 2}{\lambda_z}$ (NOTE: $\lambda_z$ is the terminal phase rate constant). |
| AUC <sub>(0-t)</sub> | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the loge trapezoidal rule for each decremental trapezoid. |
| AUC <sub>(0-∞)</sub> | Area under the concentration-time curve extrapolated to infinity will be calculated (after single dose only) as: $AUC_{(0-\infty)} = AUC_{(0-t)} + C(t)/\lambda_z$ (NOTE: $\lambda_z$ is the terminal phase rate constant). |
| %AUC <sub>ex</sub> | [The percentage of $AUC_{(0-\infty)}$ obtained by extrapolation (%AUC <sub>ex</sub> ) will be calculated as: $[AUC_{(0-\infty)} - AUC_{(0-t)}] / AUC_{(0-\infty)} \times 100$ |
| CL/F | Apparent Clearance |

NOTES:

Additional parameters may be included as required.

#### 8.1.2. Summary Measure

- All the derived PK parameters will be summarized through descriptive statistics.
- Part 1 (single dose): AUC<sub>(0-t)</sub>, AUC<sub>(0-\infty)</sub>, %AUC<sub>ex</sub>, t<sub>max</sub>, t<sub>lag</sub>, t<sub>1/2</sub>, C<sub>max</sub>, C<sub>last</sub>, t<sub>last</sub>, CL/F

#### 8.1.3. Population of Interest

These descriptive summaries will be based on the PK population.

#### 8.1.4. Strategy for Intercurrent (Post-Randomization) Events

Only completely administered doses of treatment will be considered for analysis. Participants may be replaced until the desired cohort size is attained. No imputation will be done for missing data after a participant withdrawal.

## 8.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Section 11.10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 8.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 8.2. Statistical Analysis of derived PK Parameters

The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).

Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

207863

#### 8.2.1. Endpoint / Variables

 $AUC_{(0-\infty)}$  and  $C_{max}$  in the single dose study part.

#### 8.2.2. Summary Measure

The summary measure will be the point estimates and 90% CIs of mean slopes of log<sub>e</sub>(dose) in the single dose study part.

#### 8.2.3. Population of Interest

The secondary pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

## 8.2.4. Strategy for Intercurrent (Post-Randomization) Events

Only completely administered doses of treatment will be considered for analysis. Analyses will be based on available PK parameters. No imputation will be done for missing PK parameters for any participant.

#### 8.2.5. Statistical Analyses / Methods

#### 8.2.5.1. Statistical Methodology Specification

- The following statistical analyses will only be performed if sufficient data is available (i.e. if subjects have well defined plasma profiles).
- Pharmacokinetic analysis will be the responsibility of the Clinical Pharmacology Modelling and Simulation Department, (CPMS) and Statistical analyses of the pharmacokinetic parameters will be the responsibility of the Biostatistics Department.

#### Pharmacokinetic Statistical Analyses - Dose Proportionality in single dose (Power Model)

#### **Endpoint / Variables**

• For SAD part: AUC<sub>(0-∞)</sub>, C<sub>max</sub>

#### **Model Specification**

Power model

$$v = \alpha * dose^{\beta}$$

where y denotes the PK parameter being analyzed and dose denotes the total dose administered to a subject.

• loge transformed data will be analyzed by fitting the following linear model:

$$log_{e}y = log_{e}\alpha + \beta log_{e}dose$$

Data from all available doses in each part of the study will be considered.

#### **Model Checking & Diagnostics**

- Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative transformations, such as data squared or square root of data, will be explored.

#### **Model Results Presentation**

Estimates of slope  $\beta$  will be reported along with corresponding 90% confidence intervals. If the CI contains 1 then we shall assume Dose Proportionality to hold.

## 9. PHARMACODYNAMIC ANALYSES

## 9.1. Pharmacodynamic Parameters and Summaries

The primary Pharmacodynamic measure is CD4 receptor occupancy (%RO) after single dose administration. Secondary measures include the component parameters of the %RO calculation and measures of activated T-cells.

#### 9.1.1. Endpoint / Variables

CD4 receptor occupancy (%RO), component parameters used to calculate %RO, and active T-cells. The parameters are measured via flow cytometry and are reported as median fluorescence intensity.

## 9.1.2. Summary Measure

The following PD parameters will be summarized descriptively by treatment at each timepoint and also as change from baseline.

| Parameter | Note |
|------------------------------------------|---------------------------|
| CD3+CD8+CD25+ (%CD8+) | Measures activated T-cell |
| CD3+CD8+ CD4(ADX6940)_AF647 MFI | Used in %RO calculation |
| CD3+CD4(OKT4)+CD25+ (%CD4(OKT4)) | Measures Activated T-cell |
| CD3+CD8- CD4(OKT4)_PE MFI | Used in %RO calculation |
| CD3+CD8- CD4(ADX6940)_AF647 MFI | Used in %RO calculation |
| CD3+CD8- CD4(ADX6940)_AF647 Adjusted MFI | |
| | Used in %RO calculation |
| % Free | Calculated % Free |
| %RO | Calculated % RO |

#### NOTE:

Additional parameters may be included as required.

2020N435833\_00 207863

# 9.1.3. Population of Interest

The primary pharmacodynamics analyses will be based on the PK population, unless otherwise specified.

# 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Since %RO is being reported descriptively, missing values will not be imputed and summaries will be based on observed data.

#### 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Section 11.10: List of Data Displays and will be based on GSK Data Standards and statistical principles.

207863 | Statistical Analysis Plan RAP 04 May 2020 | TMF-1766872 | 2.0

CONFIDENTIAL

2020N435833\_00 207863

# 10. REFERENCES

• Whitehead J. et al., Easy-to-implement Bayesian methods for dose-escalation studies in healthy participants, Biostatistics, 2, 47cs, 2, 47v 2001

2020N435833\_00 207863

# 11. APPENDICES

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

N/A as per-protocol population is not defined as an analysis population.

# 11.2. Appendix 2: Schedule of Activities

The following is the protocol-defined Schedule of Activities pertaining the Part 1 of the study.

Table 2 SCREENING AND FOLLOW-UP/EARLY DISCONTINUATION ASSESSMENTS (Part 1 and Part 2)

| | | Follow- | Notes |
|---|---|---|---|
| | Screening | up/Early | Follow-up Visit to occur approximately 28 days after last study |
| Procedure | (up to 30 days prior | Discon<br>Visit (~28 | drug administration or 5 half-lives (as determined from Part 1 |
| | to Day 1) 1 | days post | PK data), whichever is longer. |
| | to Day 1) | last dose) | |
| Outpatient Visit | Х | X | |
| Informed Consent | Х | | |
| Inclusion and Exclusion | Х | | |
| Criteria | | | |
| Demography | Х | | |
| Medical History | Х | | |
| Full Physical Examination | | | |
| (Including Height and | Χ | | Additional examinations may be performed, or brief |
| Weight at the screening | | | examinations made full examinations, by the Investigator, as |
| visit) | | | deemed necessary (e.g. where safety or laboratory findings |
| Target/Brief Physical Examination | | Χ | indicate). |
| | V | | |
| 12-lead ECG | X | X | Triplicate ECGs will be used to determine participant |
| Vital signs | X | | eligibility at screening. |
| Urine Drug Screen Alcohol Screen | X | | Additional tests may be performed by the Investigator, as deemed necessary (e.g. where safety or laboratory |
| Cotinine Screen | X | | findings indicate). Tests will be conducted within site |
| Pregnancy Test | X | X | specified standards. |
| HIV, Hep B and Hep C | ^ | ^ | specified standards. |
| Screen | Х | | |
| Tuberculosis Test | Х | | |
| Laboratory assessments | Χ | Х | |
| Pharmacokinetic sample | | Х | |
| Pharmacodynamic sample | | Х | |
| Anti- GSK3732394<br>antibodies | | Х | |
| Adverse Event Review | Х | Х | The collection of SAEs will be from the screening visit to the end of the study |

| | Screening | Follow-up/Early | Notes |
|---|---|---|---|
| Procedure | (up to 30 days<br>prior to Day 1) 1 | Discon Visit<br>(~28 days post<br>last dose) | Follow-up Visit to occur approximately 28 days after last study drug administration or 5 half-lives (as determined from Part 1 PK data), whichever is longer. |
| Concomitant Medication Review | Χ | X | |

<sup>1.</sup> Screening must be performed within 30 days prior to receiving the dose of GSK3732394/PBO on Day 1

Table 3 Part 1 - All Cohorts Inpatient Days -1 to Day 14

| | | | | | | | | | | | D | ay | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Due en desse | | | | | Day | <i>i</i> 1 | | | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Procedure | Day<br>-1 | Pre-<br>dose | 0 h | 0.5 h | 1 h | 2 h | 4 h | 8 h | 12h | 24h | 48h | 72h | 96h | 120h | 144h | 168h | 192h | 216h | 240h | 264h | 288h | 312h |
| Admission to Unit | Χ | | | • | | | - | - | | • | • | | - | - | - | • | - | • | | - | | |
| Discharge from Unit | | | | | | | | | | | | | | | | | | | | | | Х |
| Urine Drug<br>Alcohol/Screen/Cotinine | Х | | | | | | | | | | | | | | | | | | | | | |
| Brief Physical Exam | Х | | | | | | | | | Х | | | | | | Х | | | | | | Χ |
| Vital signs | | Х | | | Х | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Χ | Х | Χ | Χ | Х |
| 12-lead ECG | | X | | | | | Х | | Х | Χ | | | | | | Х | | | | | | Х |
| Pregnancy Test | Х | | | | | | | | | | | | | | | | | | | | | |
| Meals | | | | | | | | | | Pe | r site us | ual prac | tice | | | | | | | | | |
| Laboratory assessments <sup>1</sup> | Х | | | | | | | | | Х | Х | | Х | | | Х | | | Χ | | | Х |
| Randomization | | Х | | | | | | | | | | | | | | | | | | | | |
| Drug administration | | | Х | | | | | | | | | | | | | | | | | | | |
| Pharmacokinetic sample <sup>2</sup> | | Х | | Χ | Χ | Χ | Х | Х | Χ | Х | Χ | Χ | Х | Χ | Χ | Х | Χ | Х | Χ | Х | Χ | Х |
| Pharmacodynamic | | Х | | Х | Х | Х | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Χ | Х | Х | Х |

| | | | | | | | | | | | | ay | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Day | y 1 | | | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Procedure | Day<br>-1 | Pre-<br>dose | 0 h | 0.5 h | 1 h | 2 h | 4 h | 8 h | 12h | 24h | 48h | 72h | 96h | 120h | 144h | 168h | 192h | 216h | 240h | 264h | 288h | 312h |
| sample <sup>2</sup> | | | | | | | | | | | | | | | | | | | | | | |
| Antidrug Antibody sample | Х | | | | | | | | | | | | | | Х | | | Х | | | | Х |
| Biomarker sample <sup>3</sup> | Х | | | | | | | | | | | | | | | | | | | | | |
| Urine sample <sup>4</sup> | Χ | | | | | ) | ( | | | | | | | | | | | | | | | |
| SAE/AE Review <sup>5</sup> | <== | | | | | | | | | | | | | | | | | | | | | |
| Con Med Review | <== | > | | | | | | | | | | | | | | | | | | | | |

- 1. Laboratory assessments include hematology (with lymphocyte subset [CD4/CD8/CD3], clinical chemistry and urinalysis.
- 2. The number of PK and PD sampling time points may be reduced/extended in subsequent dosing groups once human PK data are available from initial SAD dosing cohorts. An aliquot of the PK serum sample will be used for GSK3732394-related material (serum metabolites) identification.
- 3. Serum for biomarkers of immune activation will be collected at baseline and post-treatment in the event of clinical symptoms
- 4. Urine will be collected at Day -1 (10mL) and for 24 hours after dose administration for GSK3732394-related material identification in the highest dose cohort only. Details for urine collection and interval is included in the SRM.
- 5. To include assessment of injection site(s) as appropriate (see also Protocol Section 3.3.1 and Protocol Section 8.1, and the SRM).

Table 4 Part 1 - Outpatient Visit Days 17, 21, 24, 28

| | | [ | Day | |
|---|---|---|---|---|
| Procedure | 17 | 21 | 24 | <b>28</b> <sup>1, 2</sup> |
| Brief Physical Exam | Х | Х | Х | Х |
| Vital signs | X | Х | X | X |
| 12-lead ECG | Х | | | Х |
| Pregnancy Test | | | | X |
| Laboratory assessments <sup>3</sup> | Х | Х | X | X |
| Pharmacokinetic sample <sup>4,5</sup> | X | Х | X | X |
| Pharmacodynamic sample <sup>4,5</sup> | X | X | X | X |
| Antidrug Antibody sample | | Х | | X |
| Biomarker sample <sup>6</sup> | | | | |
| Adverse Event Review <sup>7</sup> | <========= | | ======================================= | ======> |
| Con Med Review | <=====>> | | | |

- 6. In the event of terminal half-life longer than predicted, PK/PD and laboratory assessments will occur every four days until an estimated 5 half-lives have elapsed
- 7. For participants with no ongoing AEs or Vital Sign/Laboratory measures of clinical concern at Day 28 Visit, these procedures and those listed in Table 2 Screening and Follow-up/Early Discontinuation" for Follow-up/Early Discontinuation Visit (~28 days post last dose) may be considered the same.
- 8. Laboratory assessments include hematology (with lymphocyte subset [CD4/CD8/CD3], clinical chemistry and urinalysis.
- 9. An aliquot of this PK serum sample will be used for GSK3732394-related material (serum metabolites) identification.
- 10. PK samples collection on Days 17, 21 and 24 are conditional on the PK assessment at up to Day 7 during the conduct of the study and may be adjusted as data become available.
- 11. Serum for biomarkers of immune activation will be collected at baseline and post-treatment in the event of clinical symptoms
- 12. To include assessment of injection site(s) as appropriate (see also Protocol Section 3.3.1 and Protocol Section 8.1, and the SRM).

Table 5 Part 2 - All Cohorts Inpatient Days -1 to Day 17

| | | | | | | | | | | | | | | Day | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Da | | | | Da | ay 1 | | | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 3 | 9 | 10 | 11 | 12 | 13 | 14 | 1 | 5 | 16 | 17 |
| | Day -1 | Pre-dose | 0 h | 0.5 h | 1 h | 2 h | 4 h | 8 h | 12h | 24h | 48h | 72h | 96h | 120h | 144h | Pre-dose | 0 h | 24h | 48h | 72h | 96h | 120h | 144h | Pre-dose | 0 h | 24h | 48h |
| Admission to Unit | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine Drug/<br>Cotinine/Alcohol Screen | Х | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Brief Physical Exam | Χ | | | | | | | | | Х | | | | | | X | | | | | | | Х | | | | |
| Vital signs | | Χ | | | Х | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | | Χ | Χ | Χ | Χ | Х | Х | Χ | | Х | Х |
| 12-lead ECG | ) | ( | | | | | Х | | Χ | Х | Χ | | | | | Х | | | | | | | | Χ | | | |
| Pregnancy Test | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Meals | | | | | | | | | | | | Pe | er site | usua | l pract | tice | | | | | | | | | | | |
| Laboratory assessments <sup>1</sup> | Χ | | | | | | | | | Х | Χ | | Χ | | | Х | | Χ | | Χ | | | | Χ | | Χ | |
| Randomization | | Χ | | | | | | | | | | | | | | | | | | | | | | | | | |
| Drug administration | | | Х | | | | | | | | | | | | | | Х | | | | | | | | Χ | | |
| Pharmacokinetic sample <sup>2</sup> | | Χ | | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | Χ | Х |
| Pharmacodynamic sample | | Χ | | Χ | Χ | Χ | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | | Χ | Χ | Χ | Х | Х | Х | Χ | | Χ | Х |
| Antidrug Antibody sample | Χ | | | | | | | | | | | | | | | Х | | | | | | | | Χ | | | |
| Biomarker sample <sup>3</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Urine sample <sup>4</sup> | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Adverse Event Review <sup>5</sup> | <= | <> | | | | | | | | | | | | | | | | | | | | | | | | | |
| Con Med Review | <= | ==== | ==== | ==== | ==== | ==== | ==== | ==== | ==== | -=== | ==== | ===== | ==== | ==== | ==== | ===== | ==== | ==== | ==== | ==== | ==== | ===== | ===== | ==== | ==== | ==== | ==> |

- 1. Laboratory assessments include hematology (with lymphocyte subset [CD4/CD8/CD3], clinical chemistry and urinalysis.
- 2. An aliquot of the PK serum sample will be used for GSK3732394-related material (serum metabolites) identification. Refer to the windows allowance agreement attached to the SRM for timing of trough samples to be drawn on non-dosing days.
- 3. Serum for biomarkers of immune activation will be collected at baseline and post-treatment in the event of clinical symptoms
- 4. Urine will be collected at Day -1 (10mL) and for 24 hours after dose administration for GSK3732394-related material identification after the 4th MAD dose. Details for urine collection and interval is included in the SRM.
- 5. To include assessment of injection site(s) as appropriate (see also Protocol Section 3.3.1 and Protocol Section 8.1, and the SRM).

2020N435833\_00 207863

# 11.3. Appendix 3: Assessment Windows

• Nominal time will be used for all analysis except PK analysis where planned and actual time will be used.

# 11.3.1. Definitions of Assessment Windows for Analyses

The visit assigned to the assessment as entered in the eCRF (nominal visit) will be used for reporting.

# 11.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 11.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| In-Patient | Study Treatment Start Date < Date ≤ Study Treatment Stop Date +14 Days |
| Out-Patient<br>Follow up | Date > Study Treatment Stop Date + 14 Days |

#### 11.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before 28 days prior to screening visit |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 11.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date plus 14 days (in-patient setting) |
| | <ul> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 14 days.</li> </ul> |
| | <ul> <li>Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date</li> <li>+ 14 days.</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 11.5. Appendix 5: Data Display Standards & Handling Conventions

#### 11.5.1. Reporting Process

| Software | Software |
|---|---|
| The currently sup | The currently supported versions of SAS software will be used. |
| Reporting Area | |
| HARP Server | US1SALX00259 |
| HARP Compound | HARP Compound Compound: GSK3732394, study: 207863, reporting effort: final_01 |
| Analysis Datasets | |
| <ul> <li>Analysis datasets<br/>Version 1.1).</li> </ul> | 7 many old databate will be disasted describing to object databatics (object to voicion o.2 a ribatin to |
| Generation of RTF Files | |
| RTF files will be of | generated for SAC. |

### 11.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - Display all numeric variables with the same number of decimal places as the collected precision.
  - Display minimum and maximum values with the same number of decimal places as the collected precision.
  - Display the mean and percentiles (e.g. median, Q1, and Q3) with one additional decimal place.
  - Display the standard deviation and standard error with two additional decimal places.
  - Within a column, align all data values or summary statistics along the decimal point.
  - The reported precision for PK concentration data will be 1 decimal place but may be altered by parameter depending on the significant digits.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.

| Reporting | for [ | Data | Listings: |
|-----------|-----------|-----------------|--------------------|
| | Reporting | Reporting for I | Reporting for Data |

- Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
- Unscheduled or unplanned readings will be presented within the subject's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables and figures.
- All unscheduled visits will be included in listings.

| <b>Descriptive Summary</b> | Descriptive Summary Statistics |
|---|---|
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

# 11.5.3. Reporting Standards for Pharmacokinetic Data

| Dharmacakinatia Can | contration Data |
|---|---|
| Pharmacokinetic Con PC Windows Non- Linear (WNL) File Descriptive Summary Statistics, Graphical Displays and Listings | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [SOP_514512]. Note : Concentration values will be imputed as per GUI_51487 Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive |
| | summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | None. All PK parameters will be derived by the CPMS Pharmacokineticist. |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to [Standards for Handling NQ Impacted PK Parameters]. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Loge-transformed data: N, n, geometric mean, 90% CI of geometric mean, standard deviation (SD) of loge transformed data and between subject geometric coefficient of variation (CVb (%)) will be reported. CVb (%) = √ (exp(SD2) – 1) * 100 [NOTE: SD = SD of loge transformed data] Parameters Not Being Loge Transformed: Tmax and T1/2. |
### 11.6. Appendix 6: Derived and Transformed Data

### 11.6.1. General

### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 11.3.1) the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

### 11.6.2. Study Population

### **Treatment Compliance**

• Treatment compliance will be evaluated by comparing randomized and actual doses of each participant in the listing.

### **Extent of Exposure**

 For the single dose portion of the study each participant receives a single dose. Therefore, no cumulative dose will be calculated per participant.

### 11.6.3. Safety

### **ECG Parameters**

### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcF is machine read, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

### **ECG Parameters**

### **Corrected QT Intervals**

- When not entered directly in the eCRF (ClinBase), corrected QT intervals by Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF will be derived as :

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

### 11.6.4. Pharmacokinetic

#### PK parameters

- The PK Population will include all subjects who undergo PK sampling and have evaluable PK assay results.
- See Section 8.1 for derived Pharmacokinetic parameters

### 11.6.5. Pharmacodynamic

### % Receptor Occupancy

CD4 Free Receptor (%Free) and CD4 Receptor Occupancy (%RO) will be calculated as follows:

$$\% Free = \begin{pmatrix} \frac{\Delta CD3^{+}CD8^{-} \ ADX6940\_AF647 \ MFI \ post \ dose}{\Delta CD3^{+}CD8^{-} \ ADX6940\_AF647 \ MFI \ pre \ dose} \\ \hline \frac{CD3^{+}CD8^{-} \ OKT4\_PE \ MFI \ post \ dose}{CD3^{+}CD8^{-} \ OKT4\_PE \ MFI \ pre \ dose} \end{pmatrix} *100$$

$$\% RO = \left(1 - \frac{\frac{\Delta CD3^{+}CD8^{-} ADX6940\_AF647 \ MFI \ post \ dose}{\Delta CD3^{+}CD8^{-} \ ADX6940\_AF647 \ MFI \ pre \ dose}}{\frac{CD3^{+}CD8^{-} \ OKT4\_PE \ MFI \ post \ dose}{CD3^{+}CD8^{-} \ OKT4\_PE \ MFI \ pre \ dose}}\right) *_{100}$$

Note: The adjusted MFI (Δ) will be used to calculate Free Receptor and Receptor Occupancy values in the AF647 channel. Delta MFI values will be calculated as follows: (CD3+CD8-CD4(ADX6940)\_AF647 MFI) - (CD3+CD8+ CD4(ADX6940)\_AF647 MFI). %Free and %RO will be in the SDTM data.

2020N435833 00 207863

### % Receptor Occupancy

### Limit of Detection (LOD) of the Receptor Occupancy Assay

The limit of detection (LOD) of the receptor occupancy assay will be calculated using the cumulative placebo data of the study. The limit of detection (LOD) will be calculated as follows. For each placebo subject the average of (3+8-647 Delta / 3+8- OKT4 PE) will be calculated across all timepoints where both measures are available. This average value will be used to calculate %RO at each timepoint i as:

%RO<sub>i</sub>=(1-(3+8-647 Delta<sub>i</sub>/3+8- OKT4 PE<sub>i</sub>)/Mean(3+8-647 Delta<sub>i</sub>/3+8- OKT4 PE<sub>i</sub>))\*100.

The subject standard deviation (SD<sub>subject</sub>) of these %RO<sub>i</sub> values will be calculated for each placebo subject and LOD<sub>subject</sub> will be calculated as:

LOD<sub>subject</sub>=Mean(%RO<sub>i</sub>)<sup>1</sup> + 3\*SD<sub>subject</sub>

The cumulative LOD will be calculated by averaging the LOD<sub>subject</sub> across all placebo subjects. Imputed %RO is defined as 0 for all timepoints where the Assay-Reported %RO is below LOD except for the timepoint immediately prior to an Assay-Reported %RO above LOD and the timepoint immediately after an Assay-Reported %RO above LOD. The imputed %RO for these timepoints will be ½ of the LOD. Assayreported %RO will be used for summaries and both assay-reported and imputed %RO will be listed.

<sup>&</sup>lt;sup>1</sup> Note: Mean(%RO<sub>i</sub>)=0 by definition using the above average adjustment

## 11.7. Appendix 7: Reporting Standards for Missing Data

## 11.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined having completed all phases of the study including the last visit and the last scheduled procedure shown in the Schedule of Activities.</li> <li>Withdrawn subjects may be replaced in the study.</li> </ul> |
| | All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits. |

## 11.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is |
| | <ul> <li>excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

## 11.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |
| Concomitant | Partial dates for any concomitant medications recorded in the CRF will be imputed |

2020N435833\_00 207863

| Element | Reporting Detail |
|---|---|
| Medications/ | using the following convention: |
| Medical<br>History | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

# 11.8. Appendix 8: Values of Potential Clinical Importance

## 11.8.1. Laboratory Values

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and<br>Adverse | The Division of AIDS (DAIDS) grading for severity of laboratory toxicities and clinical adverse events, version 2.1, July 2017 will be used to assign grades to laboratory values. |
| Events | <ul> <li>When deriving the Grading for severity of laboratory toxicity only numeric<br/>criteria are considered. The following note will be included in the listing<br/>including laboratory severity output: "Grades were derived based on numeric<br/>criteria as defined in DAIDS Version 2.1 and did not take into consideration of<br/>clinical signs or symptoms which is needed for the final grade associated with<br/>the adverse event."</li> </ul> |
| | Reference ranges for all laboratory parameters collected throughout the study are provided by the laboratory. A laboratory value that is outside the reference range is considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Note: a high abnormal or low abnormal laboratory value is not necessarily of clinical concern. The laboratory reference ranges will be provided on the listings of laboratory data. Clinical laboratory test results outside of the reference range will be flagged in the listings. |

## 11.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|----------------------------|-------|------------------------|-------|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | | 450 |
| Absolute PR Interval | msec | 110 | 220 |
| Absolute QRS Interval | msec | 75 | 110 |
| QTc Interval (Bazett) | msec | | 450 |
| QTc Interval (Fridericia) | msec | | 450 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | 60 |

## 11.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | 85 | 160 |
| Diastolic Blood Pressure | mmHg | 45 | 100 |
| Heart Rate | bpm | 40 | 110 |

# 11.9. Appendix 9: Abbreviations & Trade Marks

## 11.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| LOD | Limit of Detection |
| MMRM | Mixed Model Repeated Measures |
| MFI | Median Fluorescence Intensity |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |

2020N435833\_00 207863

| Abbreviation | Description |
|---|---|
| RAMOS | Randomization & Medication Ordering System |
| RO | Receptor Occupancy |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Tmax | Time Taken to Maximum Observed Plasma Drug Concentration |
| Tlag | Lag time before observation of drug concentrations |
| t1/2 | Terminal phase half-life |
| tau | Dosing interval |
| Cmax | Maximum observed concentration |
| Ctau | Trough concentration |
| Clast | last observable concentration |
| tlast | time of last quantifiable concentration |
| AUC | Area under the concentration-time curve |
| CL/F | Apparent Clearance |
| NOAEL | No Observed Adverse Effect Level |
| DAIDS | Division of AIDS |

## 11.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| SAS |
| WinNonlin |

## 11.10. Appendix 10: List of Data Displays

## 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|------------|
| Study Population | 1.1 to 1.3 | NA |
| Safety | 3.1 to 3.17 | NA |
| Pharmacokinetic | 4.1 to 4.3 | 4.1 to 4.3 |
| Pharmacodynamic | 6.1 to 6.2 | NA |
| Section | Listings | |
| ICH Listings | 1 to 25 | |
| Other Listings | 26 to 29 | |

## 11.10.2. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

2020N435833\_00 207863

# 11.10.3. Study Population Tables

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population IDSL / Example Shell | | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | • |
| 1.1. | Safety | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | Safety | ES4 | Summary of Subject Disposition at Each Study Epoch | ICH E3 | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC |
| Protoc | ol Deviation | L | | | |
| 1.4. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC |
| Popula | ation Analysed | | | | • |
| 1.5. | Screened | SP1 | Summary of Study Populations | IDSL | SAC |
| Demog | graphic and Bas | seline Characteris | tics | • | • |
| 1.6. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC |
| 1.7. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

2020N435833\_00 207863

# 11.10.4. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | Adverse Events (AEs) | | | | |
| 3.1. | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | Safety | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT | SAC |
| Labora | tory: Chemistry | / | | , | |
| 3.3. | Safety | LB1 | Summary of Clinical Chemistry Data | | SAC |
| 3.4. | Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | | SAC |
| 3.5. | Safety | LB16 | Summary of Worst Case Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Labora | tory: Hematolo | gy | | | |
| 3.6. | Safety | LB1 | Summary of Hematology Data | | SAC |
| 3.7. | Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC |
| 3.8. | Safety | LB16 | Summary of Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline | ICH E3 | SAC |
| Labora | Laboratory: Urinalysis | | | | |
| 3.9. | Safety | UR1 | Summary of Urine Data | | SAC |
| 3.10. | Safety | UR1 | Summary of Worst Case Urinalysis Results (Discrete or Character Values) Post-Baseline Relative to Baseline | ICH E3 | SAC |

2020N435833\_00 207863

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| ECG | | | | | • |
| 3.11. | Safety | EG2 | Summary of ECG Values | | SAC |
| 3.12. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC |
| 3.13. | Safety | EG11 | Summary of Increase in QTc Values Post-Baseline Relative to Baseline by visit and Category | Add Visit Column before category. Replace "Maximum" in shell program with summary per visit. Use the following categories: • <=10ms • >10ms-20ms • >20-30ms • >30-60ms • >60ms | SAC |
| 3.14. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC |
| Vital Si | gns | | | | |
| 3.15. | Safety | VS1 | Summary of Vital Signs | | SAC |
| 3.16. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC |
| 3.17. | Safety | VS7 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | IDSL | SAC |

2020N435833\_00 207863

## 11.10.5. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | PK Concentration | | | | |
| 4.1. | PK | PK01 | Summary of GSK3732394 Plasma PK Concentration-<br>Time Data by Treatment | | SAC |
| PK Para | meters | | | | |
| 4.2. | PK | PK06 | Summary of Derived GSK3732394 Plasma Pharmacokinetic Parameters (non-transformed and log-transformed) by Treatment | | SAC |
| PK Statistical Analysis Table | | | | | |
| 4.3. | PK | mid207187<br>Table 4.4 | Summary Results of Single Dose Proportionality Assessment Using Power Model | (reference study<br>mid207187 Table 4.4) | SAC |

2020N435833\_00 207863

# 11.10.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 4.1. | PK | PK16a | Individual GSK3732394 Plasma Concentration-Time Plots (Linear and Semi-Log) by Treatment | Overlay all individual profiles per treatment in a plot. Separate plots by treatment. | SAC |
| 4.2. | PK | PK17 | Median GSK3732394 Plasma Concentration-Time Plots (Linear and Semi-Log) | | SAC |
| 4.3. | PK | PK18 | Mean GSK3732394 Plasma Concentration-Time Plots (Linear and Semi-Log) | | SAC |

## 11.10.7. Pharmacodynamic Tables

| Pharma | Pharmacodynamic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PD | | | | | |
| 6.1. | PK | LB1 | Summary of Pharmacodynamic Parameters by Treatment | | SAC |
| 6.2. | PK | LB1 | Summary of Pharmacodynamic Parameters Changes from Baseline by Treatment | | SAC |

2020N435833\_00 207863

# 11.10.8. ICH Listings

| ICH: List | ings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject I | Disposition | | | · | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | Screened | ES9 | Listing of Subjects Who Were Rescreened | | SAC |
| 3. | Safety | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 4. | Safety | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | Safety | TA1 | Listing of Randomized and Actual Treatment | IDSL | SAC |
| Protocol | Deviations | | | | |
| 6. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Demogra | aphic and Baseline C | haracteristics | | | |
| 8. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC |
| 9. | Safety | DM9 | Listing of Race | ICH E3 | SAC |
| Concom | itant Medications | | | | |
| 10. | Safety | CM3 | Listing of Concomitant Medications | IDSL | SAC |
| Exposur | е | | | , | • |
| 11. | Safety | EX3 | Listing of Exposure Data | ICH E3 | SAC |
| Adverse | Events | | | | |

2020N435833\_00 207863

| ICH: Lis | tings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 12. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 13. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC |
| Serious | and Other Significan | t Adverse Events | | | |
| 14. | Safety | AE8CPA | Listing of Serious Adverse Events (Fatal & Non-Fatal) | ICH E3 | SAC |
| 15. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | ICH E3 | SAC |
| Hepatob | piliary (Liver) | | | | |
| 16. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL | SAC |
| 17. | Safety | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory<br>Criteria Post-Baseline | IDSL | SAC |
| 18. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | IDSL | SAC |
| 19. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | IDSL list available substance use data for subjects with liver events | SAC |
| All Labo | oratory | | | | |
| 20. | Safety | LB5A | Listing of All Laboratory Data | ICH E3 | SAC |
| ECG | | | | | |
| 21. | Safety | EG3 | Listing of All ECG Values | | SAC |

2020N435833\_00 207863

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 22. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC |
| 23. | Safety | EG5 | Listing of All ECG Findings | | SAC |
| Vital Sig | jns | | | | |
| 24. | Safety | VS4 | Listing of All Vital Signs | | SAC |
| 25. | Safety | VS4 | Listing of All Vital Signs for Subjects with Values of Potential Clinical Importance | | SAC |

# 11.10.9. Non-ICH Listings

| Non-ICH | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 26. | PK | PK07 | Listing of GSK3732394 Plasma PK Concentration-Time Data | | SAC |
| 27. | PK | PK13 | Listing of Derived GSK3732394 Plasma PK Parameters | | SAC |
| PD | | | | | |
| 28. | PK | PK07 | Listing of Assay-Reported and Imputed %Receptor Occupancy | Replace Concentration in Example Shell with %RO and add Column for Imputed %RO | SAC |
| Immuno | Immunogenicity | | | | |
| 29. | PK | IMM2 | Listing of Immunogenicity Results | | SAC |